CLINICAL TRIAL: NCT01025947
Title: Observational Study on Cryptogenic Stroke and Atrial Fibrillation Detection Through Implantable Loop Recorder
Brief Title: "Cryptogenic Stroke and Atrial Fibrillation Detection Through Implantable Loop Recorder (ILR)"
Acronym: CRYPTONITE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Collaborators: Hospital Universitario Virgen de la Arrixaca (Other); Universidad de Murcia (Other)
Responsible Party: Ricardo Ruiz Granell, MD, PhD, Hospital Clínico Universitario de Valencia
Other Study IDs: HCUV
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Atrial fibrillation; Cryptogenic stroke; Implantable loop recorder
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Patients with cryptogenic stroke (TOAST criteria) and with an implantable EKG loop recorder implanted

SUMMARY:
STUDY TYPE:

Prospective, national , multicenter, and observational study.

OBJECTIVE:

To assess the incidence of AF in patients with cryptogenic stroke who have implanted an AF detection device during a period of 2 years.

DEVICE:

Reveal XT 9529 (SQDM)

SAMPLE SIZE AND STUDY DURATION:

100 patients enrolled which will be followed during a period of 2 years.

DETAILED DESCRIPTION:
Observational study in patients with cryptogenic stroke (TOAST criteria) and with an implanted EKG loop recorder, with the primary objective of knowing the atrial fibrillation incidence in this population

ELIGIBILITY:
Inclusion Criteria:

* All patients included must meet one of these two conditions:

  * Patient presenting with an episode of transient ischemic attack (TIA) of cryptogenic origin with neurological symptoms of less than 24h of evolution and negative neuroimaging.
  * First episode of ischaemic stroke with cryptogenic etiology following TOAST criteria
* All patients must meet all of the following:

  * The patient has been implanted an ILR within 30 days after qualifying event
  * Age between 45-85 years
  * No stenosis >50% in any arterial vessel corresponding to the affected territory
  * Normal Echocardiography
  * Normal 24 hours EKG Holter recording
  * Absence of Patent Foramen Ovale through transcranial doppler (or transesophageal echocardiography)
  * Acceptance and signature of Patient Informed Consent.

Exclusion Criteria:

* All patients included cannot meet any of the following conditions:

  * Recurrent stroke or TIA
  * Stroke or TIA with determined etiology according to TOAST criteria.
  * Anticoagulation indication at the time of enrollment in the study.
  * Total contraindication for anticoagulation therapy
  * Atrial fibrillation detection prior to enrollment
  * Severe cognitive impairment or dementia
  * Patient unable to be followed up
  * Patients enrolled in another clinical trial
  * Patients with life expectancy of less than 1 year
  * Pregnancy

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cryptogenic stroke (TOAST criteria) and with an implantable EKG loop recorder implanted for detection of atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
First AF episode detected by the implantable loop recorder in patients that had a cryptogenic stroke. An AF episode will be considered an AF episode that lasts at least 2 minutes. | Patients will be followed up during two years, regardless of reaching or not the primary endpoint.

SECONDARY OUTCOMES:
All subsequent AF episodes detected by the ILR after primary outcome (AF burden) | Patients will be followed up during two years
AF episodes detected by external monitoring | Patients will be followed up during two years
Presence of stroke, recurrent TIA, or silent infarction in neuroimaging | Patients will be followed up during two years
Changes in anticoagulant therapy | Patients will be followed up during two years

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Ruiz-Granell, MD, Phd, Principal Investigator — Hospital Clinico Universitario de Valencia; Arcadio Garcia-Alberola, MD, PhD, Study Chair — Hospital Universitario Virgen de la Arrixaca; Ana Morales, MD, Study Chair — Hospital Universitario Virgen de la Arrixaca; Alejandro Ponz, MD, Study Chair — Hospital Clinico Universitario de Valencia
Locations (2):
- Spain (2):
  - Hospital Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia

REFERENCES:
- [Background] Rosamond W, Flegal K, Friday G, Furie K, Go A, Greenlund K, Haase N, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell CJ, Roger V, Rumsfeld J, Sorlie P, Steinberger J, Thom T, Wasserthiel-Smoller S, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2007 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2007 Feb 6;115(5):e69-171. doi: 10.1161/CIRCULATIONAHA.106.179918. Epub 2006 Dec 28. No abstract available. PMID 17194875
- [Background] Carandang R, Seshadri S, Beiser A, Kelly-Hayes M, Kase CS, Kannel WB, Wolf PA. Trends in incidence, lifetime risk, severity, and 30-day mortality of stroke over the past 50 years. JAMA. 2006 Dec 27;296(24):2939-46. doi: 10.1001/jama.296.24.2939. PMID 17190894
- [Background] Adams HP Jr, Bendixen BH, Kappelle LJ, Biller J, Love BB, Gordon DL, Marsh EE 3rd. Classification of subtype of acute ischemic stroke. Definitions for use in a multicenter clinical trial. TOAST. Trial of Org 10172 in Acute Stroke Treatment. Stroke. 1993 Jan;24(1):35-41. doi: 10.1161/01.str.24.1.35. PMID 7678184
- [Background] Adams HP Jr, Davis PH, Leira EC, Chang KC, Bendixen BH, Clarke WR, Woolson RF, Hansen MD. Baseline NIH Stroke Scale score strongly predicts outcome after stroke: A report of the Trial of Org 10172 in Acute Stroke Treatment (TOAST). Neurology. 1999 Jul 13;53(1):126-31. doi: 10.1212/wnl.53.1.126. PMID 10408548
- [Background] Sacco RL, Ellenberg JH, Mohr JP, Tatemichi TK, Hier DB, Price TR, Wolf PA. Infarcts of undetermined cause: the NINCDS Stroke Data Bank. Ann Neurol. 1989 Apr;25(4):382-90. doi: 10.1002/ana.410250410. PMID 2712533
- [Background] Jabaudon D, Sztajzel J, Sievert K, Landis T, Sztajzel R. Usefulness of ambulatory 7-day ECG monitoring for the detection of atrial fibrillation and flutter after acute stroke and transient ischemic attack. Stroke. 2004 Jul;35(7):1647-51. doi: 10.1161/01.STR.0000131269.69502.d9. Epub 2004 May 20. PMID 15155965
- [Background] Douen AG, Pageau N, Medic S. Serial electrocardiographic assessments significantly improve detection of atrial fibrillation 2.6-fold in patients with acute stroke. Stroke. 2008 Feb;39(2):480-2. doi: 10.1161/STROKEAHA.107.492595. Epub 2008 Jan 3. PMID 18174488
- [Background] Liao J, Khalid Z, Scallan C, Morillo C, O'Donnell M. Noninvasive cardiac monitoring for detecting paroxysmal atrial fibrillation or flutter after acute ischemic stroke: a systematic review. Stroke. 2007 Nov;38(11):2935-40. doi: 10.1161/STROKEAHA.106.478685. Epub 2007 Sep 27. PMID 17901394
- [Background] Solano A, Menozzi C, Maggi R, Donateo P, Bottoni N, Lolli G, Tomasi C, Croci F, Oddone D, Puggioni E, Brignole M. Incidence, diagnostic yield and safety of the implantable loop-recorder to detect the mechanism of syncope in patients with and without structural heart disease. Eur Heart J. 2004 Jul;25(13):1116-9. doi: 10.1016/j.ehj.2004.05.013. PMID 15231369